CLINICAL TRIAL: NCT05680870
Title: The Possible Protective Role of Omeprazole Against Oxaliplatin Induced Neuropathy in Patients With Cancer Treated With Oxaliplatin-fluorouracil Chemotherapy Protocols
Brief Title: The Possible Protective Role of Omeprazole Against Oxaliplatin Induced Neuropathy in Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aya Mohamed Sadek Elsaid (Other)
Responsible Party: Sponsor-Investigator, Aya Mohamed Sadek Elsaid, Clinical phatmacist, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MS.22.12.2244.R1
Record Dates: First submitted 2022-12-28; First posted 2023-01-11 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy
Keywords: Peripheral neuropathy; Colorectal cancer; Pancreatic cancer
MeSH Terms: conditions — Peripheral Nervous System Diseases; Colorectal Neoplasms; Pancreatic Neoplasms | interventions — Omeprazole

STUDY DESIGN:
Intervention Model Description: 46 participants will be classified into 2 arms : intervention arm will receive omeprazole plus chemotherapy Control arm will receive chemotherapy only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Control grp will not receive omeprazole . They will receive chemotherapy protocols only
- Intervention group (Experimental): Intervention group will receive omeprazole plus chemotherapy protocols
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole — Omeprazole 40 mg 3 times daily for 5 days ..to start 2 days before chemotherapy cycles
  Other Names: Omez
  Arms: Intervention group

SUMMARY:
Oxaliplatin(OXA) chemotherapy protocols are used in treatment of cancers like colorectal (CRC) and pancreatic cancer. OXA causes peripheral neuropathy which is considered treatment limiting factor. In recent studies, it shows that omeprazole(OME) has antioxidant effect and can inhibit organic cation transporter 2 (OCT2) in kidney. So OME can protect against peripheral neuropathy induced by OXA through oxidative stress . Also OME activates extracellular-signal-regulated kinase(ERK) / mitogen activated protein kinase ( MAPK) pathway, so improves demyelinating symptoms.

DETAILED DESCRIPTION:
Randomized controlled parallel study

Forty-six patients with pancreatic cancer or CRC who receive OXA 85mg/m2 in their protocols scheduled as a cycle every two consecutive weeks for 6 months to receive 12 cycles. Patients will be recruited from Clinical Oncology and Nuclear Medicine Department, Mansoura University Hospital, Mansoura, Egypt. The patients will be randomized using sealed envelope method into two groups:

According to the results of previous studies, the total number of subjects required detecting the effect of neuro-protective drugs in patients received chemotherapy with 5% significance and 80% power and attrition rate equal to 15% was 41 . In this context, during the current study, a total sample size 42 patients in both arms will be sufficient to provide a good power to detect the effect. Assuming that the attrition rate will be 10% the initial sample size will be 46 patients in both arms.

Assessment of patient adherence and evaluation of drug safety The medication will be provided on biweekly intervals and the participants adherence will be assessed through counting the pills and by medications refilling rate. Participants will also followed-up by telephone calls and through direct meetings during chemotherapy cycles to assess their adherence and report any drugs related adverse effects using adverse drug reactions reporting form the adverse effects will be also collected through patients' laboratory data and patient sheet. The patients will be asked about any adverse effects related to study medication. Patients will be considered non-adherent and excluded from the study if consumed less than 90% of study medication at any month of the study duration.

Statistical analysis - Statistical analysis will be done by the statistical software package version 25 . Data will be tested for normality using Kolmogorov-Smirnov and Shapiro wilk tests. Normally distributed data will be analyzed using paired and un-paired t-test. Non normally distributed data will be compared using Mann-Whitney U test. Also, Mann-Whitney U test will be used to compare non-parametric data between the two arms including the neuropathy grading and the Neurotoxicity-12(NTX-12) total scores. Categorical data will be computed by Chi-square test. - Fisher exact test will be used to analyze the reported adverse effects. - Correlation between variables will be analyzed by Pearson or spearman correlation what appropriate. - The significance level was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnose cases with colorectal (CRC)and pancreatic cancers (males and females) ≥ 18 years old, and ≤ 65 years old.
* Patients who will scheduled to receive modified FOLFOX-4,6,7 (OXA, Leucovorin, and 5-fluorouracil) or mFOLFIRINOX (OXA, irinotecan,leucovorin, and 5-Fluorouracil) for 12 cycles.
* Patients with performance status 0-2 according to Eastern Cooperative Oncology Group (ECOG) Score.

Exclusion Criteria:

* Evidence of pre-existing peripheral neuropathy resulting from another reason (documented patients with brain tumor, brain trauma, seizures or any other neuropathic disorder).
* CRC patients receiving protocols containing capecitabine.
* Diabetic patients.
* Documented Patients with lupus (SLE), or any other autoimmune disease.
* Documented Patients with osteoporosis or fractures.
* Prior exposure to neurotoxic chemotherapy for at least 6 months prior to the study.
* Concomitant use of other neuroprotective medications (gabapentin, lamotrigine, phenytoin, tricyclic antidepressants, etc.,).
* Patients taking medications that omeprazole can interact with or affect their metabolism, such as (digoxin, ketoconazole, methotrexate, clopidogrel, marevan, etc.,).
* Pregnant and breastfeeding women.
* Patients with abnormal renal function (S.cr > 1.5 mg/dl or crcl < 45 ml/min).
* Patients with liver diseases (serum bilirubin > 1.5 mg/dl / Alanine transaminase, Aspartate transaminase > 2-4 ULN).
* Smokers or documented patients with condition associated with oxidative stress.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Acute peripheral neuropathy | After the first intervention by 2 weeks of the first chemotherapy cycle ( each cycle is two days every two weeks), and through the study average for six months
  the percentage of patients with acute peripheral sensory neuropathy grade ≥ 2 and the variation of both 12-item neurotoxicity questionnaire (Ntx-12) total score and pain rating scale score
Chronic peripheral neuropathy | After the end of 12 chemotherapy cycles ( after six months of interventions)
  Percentage of patients who have developed chronic peripheral neuropathy grade ≥ 2 after the end of 12 cycles and the variation of both NTX-12 total score and pain rating scale

SECONDARY OUTCOMES:
Malonaldehyde | After 3 months of treatment
  Changes in malonaldehyde level
Neurotensin | After 3 months of treatment
  Changes in neurotensin level
OCT | After 3 months of treatment
  Changes in OCT level

CONTACTS AND LOCATIONS:
Overall Officials: Sahar K Hegazy, Professor, Study Director — Professor of clinical pharmacy , faculty of pharmacy, Tanta university
Locations (1):
- Tanta university, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No